CLINICAL TRIAL: NCT02628847
Title: Sildenafil and Stroke Recovery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment was problematic
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lorie Richards, Chair and Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 53515
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; motor skills; sildenafil citrate; White matter
MeSH Terms: conditions — Stroke | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): Sildenafil citrate 25mg once per day for 14 days starting day 5-9 post stroke while undergoing usual rehabilitation
  Interventions: Drug: sildenafil citrate
- control (Placebo Comparator): placebo capsule once per day for 14 days starting day 5-9 post stroke while undergoing usual rehabilitation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sildenafil citrate
  Other Names: Viagra
  Arms: Drug
Drug: Placebo
  Arms: control

SUMMARY:
This is a small, pilot randomized clinical trial of administering sildenafil citrate to individuals within 10 days of ischemic stroke who have motor impairment and who are undergoing inpatient rehabilitation compared to placebo. The primary outcome is motor recovery at one and three months.

DETAILED DESCRIPTION:
Individuals who are within 4-10 days post ischemic stroke with arm hemiparesis or hemiplegia who are admitted to inpatient rehabilitation are randomized to receive either sildenafil citrate (25 mg once per day) or placebo for 14 days. These individuals receive usual rehabilitation and medical care. Primary outcomes are motor skills and walking speed at one and three months.

If willing and able, participants undergo an MRI to measure the integrity of the white matter pathways in the motor system using diffusion tensor imaging. Repeat MRIs are obtained at one and three months. The investigators will examine if such white matter integrity predicts response to the drug and if the drug facilitates changes in white matter.

ELIGIBILITY:
Inclusion Criteria:

1. between 4 and 9 days post-ischemic stroke;
2. admitted to inpatient rehabilitation;
3. cognitively able to provide consent or assent;
4. were living independently in the community prior to their stroke.

Exclusion Criteria:

1. hemorrhagic stroke or subarachnoid hemorrhage;
2. other neurological or psychiatric conditions deemed by the investigator to impair participation;
3. no previous stroke on same side of brain unless that stroke was cerebellar
4. moribound or not expected to live 6 months;
5. contraindications to taking sildenafil in pill or syrup form;
6. other medical conditions that would limit ability to participate in the study, specifically a) currently taking the P450 enzyme inhibitors (erythromycin, ketoconazole, itraconazole, saquinavir), b) currently taking the protease inhibitor ritonavir, c) currently taking nitrates or have a history of requiring nitrates treatment, d) have left ventricular outflow obstruction (i.e., aortic stenosis, idiopathic hypertrophic subaortic stenosis as confirmed by review of standard of care echo received before admission to rehabilitation), e) have severely impaired autonomic control of blood pressure, f) have previous history of symptomatic hypotension, g) have severely impaired hepatic function, h) is pregnant or become pregnant during the course of the study, i) Any medical condition which, in the opinion of the investigator, may compromise compliance with the objectives and/or procedures of the protocol.
7. scores > 50 on the upper extremity section of the Fugl-Meyer or no walking/gait impairment

   For the MRI portion of the study only:
8. contraindication to MRI: ferrous metal in body, lead included body art, claustrophobia, pacemaker
9. allergic to or had previous reaction to gadolinium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Assessment | change from baseline at 1 month
  An assessment of upper extremity and lower extremity motor impairment
Fugl-Meyer Assessment | change from baseline at 3 months
  An assessment of upper extremity and lower extremity motor impairment

SECONDARY OUTCOMES:
10 meter walk | change from baseline at one month
  an assessment of usual gait speed
Wolf Motor Function Test | baseline, one month, three months
  An assessment of motor function
Motor Activity Log | one month
  A self-report of paretic arm (frequency and perceived ability) use in every day activities
Stroke Impact Scale | one month
  A self-report measure of the impact of stroke on the individual for body functions, activities, and participation
10 meter walk | change from baseline at 3 months
  an assessment of usual gait speed
Wolf Motor Function Test | change from baseline at 3 months
  An assessment of motor function
Motor Activity Log | 3 months
  A self-report of paretic arm (frequency and perceived ability) use in every day
Stroke Impact Scale | 3 months
  A self-report measure of the impact of stroke on the individual for body

OTHER OUTCOMES:
Number of participants with unsafe Blood pressure change | one month
  blood pressure reductions or increases while taking the drug/placebo
number of participants with cardiovascular side effects | one month
  cardiovascular events, such as heart attack, angina pectoris, heart failure
number of participants with visual side effects | one month
  new abnormal color vision, light sensitivity, blurred vision or other visual side effects
number of participants with auditory or vestibular side effects | one month
  new loss of hearing, tinnitus, dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Lorie G Richards, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang RL, Chopp M, Roberts C, Wei M, Wang X, Liu X, Lu M, Zhang ZG. Sildenafil enhances neurogenesis and oligodendrogenesis in ischemic brain of middle-aged mouse. PLoS One. 2012;7(10):e48141. doi: 10.1371/journal.pone.0048141. Epub 2012 Oct 31. PMID 23118941
- [Result] Zhang L, Zhang RL, Wang Y, Zhang C, Zhang ZG, Meng H, Chopp M. Functional recovery in aged and young rats after embolic stroke: treatment with a phosphodiesterase type 5 inhibitor. Stroke. 2005 Apr;36(4):847-52. doi: 10.1161/01.STR.0000158923.19956.73. Epub 2005 Mar 3. PMID 15746452
- [Result] Zhang R, Wang Y, Zhang L, Zhang Z, Tsang W, Lu M, Zhang L, Chopp M. Sildenafil (Viagra) induces neurogenesis and promotes functional recovery after stroke in rats. Stroke. 2002 Nov;33(11):2675-80. doi: 10.1161/01.str.0000034399.95249.59. PMID 12411660
- [Result] Li L, Jiang Q, Zhang L, Ding G, Gang Zhang Z, Li Q, Ewing JR, Lu M, Panda S, Ledbetter KA, Whitton PA, Chopp M. Angiogenesis and improved cerebral blood flow in the ischemic boundary area detected by MRI after administration of sildenafil to rats with embolic stroke. Brain Res. 2007 Feb 9;1132(1):185-92. doi: 10.1016/j.brainres.2006.10.098. Epub 2006 Dec 26. PMID 17188664
- [Result] Ding G, Jiang Q, Li L, Zhang L, Zhang ZG, Ledbetter KA, Gollapalli L, Panda S, Li Q, Ewing JR, Chopp M. Angiogenesis detected after embolic stroke in rat brain using magnetic resonance T2*WI. Stroke. 2008 May;39(5):1563-8. doi: 10.1161/STROKEAHA.107.502146. Epub 2008 Mar 20. PMID 18356548
- [Result] Ding G, Jiang Q, Li L, Zhang L, Zhang ZG, Ledbetter KA, Panda S, Davarani SP, Athiraman H, Li Q, Ewing JR, Chopp M. Magnetic resonance imaging investigation of axonal remodeling and angiogenesis after embolic stroke in sildenafil-treated rats. J Cereb Blood Flow Metab. 2008 Aug;28(8):1440-8. doi: 10.1038/jcbfm.2008.33. Epub 2008 Apr 16. PMID 18418368
- [Result] Ding G, Jiang Q, Li L, Zhang L, Zhang Z, Lu M, Li Q, Gu S, Ewing J, Chopp M. Longitudinal magnetic resonance imaging of sildenafil treatment of embolic stroke in aged rats. Stroke. 2011 Dec;42(12):3537-41. doi: 10.1161/STROKEAHA.111.622092. Epub 2011 Sep 8. PMID 21903952
- [Result] Silver B, McCarthy S, Lu M, Mitsias P, Russman AN, Katramados A, Morris DC, Lewandowski CA, Chopp M. Sildenafil treatment of subacute ischemic stroke: a safety study at 25-mg daily for 2 weeks. J Stroke Cerebrovasc Dis. 2009 Sep-Oct;18(5):381-3. doi: 10.1016/j.jstrokecerebrovasdis.2009.01.007. PMID 19717023